CLINICAL TRIAL: NCT02865746
Title: Periapical Injection of Betamethasone to Control Postoperative Pain in Emergency Endodontic Care - A Randomized Double Blind Clinical Trial
Brief Title: Betamethasone to Control Postoperative Pain in Emergency Endodontic Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ufvjm
Record Dates: First submitted 2016-08-01; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Pain
Keywords: Steroids; Pain measurement
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group betamethasone (Active Comparator): Active Comparator: betamethasone disodium phosphate at a concentration of 4 mg / ml - dosage of 0.05 mg / kg
  Interventions: Drug: Bethametasone
- Group placebo (Placebo Comparator): sterile saline solution (sodium chloride 0.9% - 1 ml ampoules) - dosage of 0.05 mg / kg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bethametasone — The injections were performed with the aid of syringes fitted with ultrafine needles (BD ultrafine U-100, 0.3 x 8 mm), in the buccal mucosa, submucosally near the tooth's periapex of the periapical region of the tooth involved, by using the submucosal infiltration technique.
  Other Names: Group 1
  Arms: Group betamethasone
Drug: Placebo — The injections were performed with the aid of syringes fitted with ultrafine needles (BD ultrafine U-100, 0.3 x 8 mm), in the buccal mucosa, submucosally near the tooth's periapex of the periapical region of the tooth involved, by using the submucosal infiltration technique.
  Other Names: Group 2
  Arms: Group placebo

SUMMARY:
The objective of this randomized double-blind study was to evaluate the effect of betamethasone in the control of postoperative pain in patients undergoing endodontic treatment.

DETAILED DESCRIPTION:
To prevent post endodontic treatment pain, systemic administration of corticosteroids may have their effect maximized if the infiltration is performed in the oral mucosa, near the periapex of the tooth, which concentrates the inflammatory process. The administration of corticosteroids at this moment, taking advantage of the anesthetic effect still present, ensures continuous comfort during the postoperative period.

The objective of this randomized double-blind clinical trial was to evaluate the effect of the systemic administration of betamethasone - through infiltration in the oral mucosa - to control pain and edemas in patients undergoing emergency endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals had to have a tooth with pain of endodontic origin justifying emergency care;
* Individuals diagnosed with irreversible pulpitis or necrosis associated to pericementitis.

Exclusion Criteria:

Individuals who presented:

* Pregnancy or lactation;
* Use of corticosteroids;
* History of hypersensitivity to the drugs used in this study;
* Pain associated with abscesses of endodontic origin;
* Individuals with tuberculosis;
* Individuals with systemic fungal infections;
* Individuals with simple ocular herpes;
* Individuals with glaucoma;
* Individuals with acute psychosis.
* Individuals with psychotic tendencies.

Ages: 10 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-07; Primary Completion 2005-05 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Pain determined using the "Point Verbal Rating Scale - Modified VRS4" | 4 hours after treatment
  During the post-surgical interval of 4 hours, the pain was determined using the "Point Verbal Rating Scale - Modified VRS4"
Pain determined using the "Point Verbal Rating Scale - Modified VRS4" | 24 hours after treatment
  During the post-surgical interval of 24 hours, the pain was determined using the "Point Verbal Rating Scale - Modified VRS4"
Pain determined using the "Point Verbal Rating Scale - Modified VRS4" | 48 hours after treatment
  During the post-surgical interval of 48 hours, the pain was determined using the "Point Verbal Rating Scale - Modified VRS4"

SECONDARY OUTCOMES:
Analgesic consumption | 4 hours after treatment
  Each patient was contacted by phone to answer how many analgesic pills have taken. None, 1, 2 or more.
Analgesic consumption | 24 hours after treatment
  Each patient was contacted by phone to answer how many analgesic pills have taken. None, 1, 2 or more.
Analgesic consumption | 48 hours after treatment
  Each patient was contacted by phone to answer how many analgesic pills have taken. None, 1, 2 or more.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos P. Pinheiro, PhD, Principal Investigator — Federal University of Valleys of Jequitinhonha and Mucuri
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided